CLINICAL TRIAL: NCT01010711
Title: Study for Documentation of the Influence of a Specific Dietary Supplement Treatment of Migraine in Children and Adolescents
Brief Title: Influence of a Dietary Supplement as Treatment of Migraine in Children and Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Complen Health GmbH (Industry)
Responsible Party: Dr. Margarete Doppler, COMPLEN HEALTH GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOM-DS-CH-1
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Migraine
Keywords: migraine; children; dietary supplement; q10; prevention
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- migraine dietary supplement (Other): the average days of migraine during a 4 week-run-in-period are compared with the average days of migraine during intervention with a "specific dietary supplement" from week 8 - 12
  Interventions: Dietary Supplement: Migra 3

INTERVENTIONS:
Dietary Supplement: Migra 3 — powder containing coenzyme q10, blueberries, black current, vitamins, magnesium,trace elements

SUMMARY:
Migraine in children and adolescents can be associated with low serum levels of coenzyme q10, the key-enzyme of mitochondrial energy production.During migraine attacks inflammation is an important issue. Based on a double-blind placebo-controlled trial with coenzyme q10 in adults it is hypothesized that daily supplementation of coenzyme q10 as well as different antioxidative phytochemicals (from berries) and specific minerals and vitamins are able to reduce the "days with migraine" as primary parameter (open clinical trial).

DETAILED DESCRIPTION:
Children or adolescents with migraine and both parents are informed in detail about the study.Probands are advised to fill in a special childrens´ diary for migraine daily. After a 4 week-run-in period they start to take the dietary supplement (powder to be dissolved in water)plus a capsule with omega-3-fatty acids from fish oil for 12 weeks daily. Afterwards there is a follow-up without supplement treatment for another 12 weeks.76 participants will be included in the trial for statistical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* at least 3 days of migraine per month

Exclusion Criteria:

* not able to communicate in german or english language
* any disease that forbids the participation in the trial according to the investigators assessment
* pregnancy
* no willingness to participate in the trial
* known allergy to fish or soya

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-12 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
number of days with headache before and after 12 weeks of daily treatment with a migraine specific dietary supplement | headaches before and after 12 weeks of treatment

SECONDARY OUTCOMES:
frequency, duration and intensity of the migraine | before and after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Charly Gaul, MD, Principal Investigator — Universiätsklinikum Essen Neurologische Klinik, Westdeutsches Kopfschmerzzentrum, Hufelandstr.26, D-45147 Essen
Locations (2):
- Germany (2):
  - Universiätsklinikum Essen Neurologische Klinik, Westdeutsches Kopfschmerzzentrum, Hufelandstr.26,, Essen, North Rhine-Westphalia
  - Migräne und Kopfschmerzklinik Königstein, Königstein im Taunus